CLINICAL TRIAL: NCT01105572
Title: Study of Impact of Home Biomonitoring With Nurse Case Manager Support for a Congestive Heart Failure Cohort, Compared to Case Manager Support Without Biomonitoring
Brief Title: Aetna_Intel Medicare Home Biomonitoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aetna, Inc. (Industry)
Collaborators: Intel Corporation (Industry)
Responsible Party: Marcia Wade, Aetna, Inc
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Biomonitoring099
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intel Home Health Guide (Experimental): Participants in the intervention group will receive the use of the Intel Healthguide, an Internet-connected device with member-customized protocols and response algorithms. Participants interact with the Intel HealthGuide device, receiving immediate feedback when transmitting blood pressure, weights and responses to questions to a site monitored by their nurse case manager. Medicare Case Managers review and coordinate services for members with multiple and complex needs with identified gaps in their care. Medicare Case Management staff strives to enhance the member's quality of life, support continuity of care, facilitate provision of services in the appropriate setting and manage cost and resource allocation to promote quality, cost-effective outcomes.
  Interventions: Device: Intel Health Guide
- Case Management Only (No Intervention): All participants in the comparison group, are identified for outreach and assistance by a nurse case manager. Specialized Medicare Case Managers review and coordinate services for members with multiple and complex needs with identified gaps in their care. Medicare Case Management staff strives to enhance the member's quality of life, support continuity of care, facilitate provision of services in the appropriate setting and manage cost and resource allocation to promote quality, cost-effective outcomes.
  Interventions: Other: Case Management

INTERVENTIONS:
Device: Intel Health Guide — An Internet-connected device with member-customized protocols and response algorithms. Participants interact with the Intel HealthGuide device, receiving immediate feedback, and also transmitting blood pressure, weights and responses to questions to a site monitored by their nurse case manager.
  Arms: Intel Home Health Guide
Other: Case Management — Specialized Medicare Case Managers review and coordinate services for members with multiple and complex needs with identified gaps in their care Medicare Case Management staff strives to enhance the member's quality of life, support continuity of care, facilitate provision of services in the appropriate setting and manage cost and resource allocation to promote quality, cost-effective outcomes. Specially trained Medicare Case Managers collaborate with the member, family, caregiver, member authorized representative, treating practitioner, health care provider, community services and other Aetna programs to coordinate care, with a focus on member education and maximizing quality outcomes.
  Arms: Case Management Only

SUMMARY:
The hypothesis is that use of Internet-connected home biomonitoring of weight, blood pressure and other indicators, in conjunction with nurse case management, will result in improved outcome for Medicare beneficiaries with with Congestive Heart Failure; compared to case management assistance without the biomonitoring device.

DETAILED DESCRIPTION:
Goals of the Study:

* Demonstrate synergy between the Intel® Health Guide home biomonitoring and nurse case management. Measure positive impact on member engagement and clinical outcomes for members with Heart Failure.
* Quantify the potential to avoid costly re-hospitalization based on the Intel® Health Guide - enhanced case management interaction through early alerts and early intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aetna Medicare (PFFS, HMO/PPO fully insured) Individual members, plus Medicare members from any plan sponsor that has agreed it would like its members to be included
* Member meets Aetna Health Profile Database criteria for Chronic Heart Failure (Disease Management Eligibility = Y) with a disease risk stratification score of 3 - 5 (moderately severe to severe). These proprietary criteria yield a group of individuals for whom historical claims data estimates a substantial risk of hospital readmission within the coming 6 months.
* Acute inpatient admission or 2 or more emergency room visits within 6 months prior to identification
* Residence in the designated geographic areas selected for the study (The planned source population is all New Jersey, New York, Pennsylvania and North Central Aetna Individual Medicare members and North Central. If members identified from these states have not filled the study within three months, the source population may be expanded to include Aetna's North Central region members in Illinois and Ohio. These North Central members would include all Aetna Medicare Individual members in these areas, plus any Group Medicare members from Groups whose Plan Sponsors agree that the study may be offered to the members.)
* Member may be currently open/ active in case management
* Responds telephonic outreach to offer study participation, or to Interactive Voice Response outreach call, and confirms each of:

  * Their own identity {secure Health Insurance Portability Accountability Act (HIPAA) compliant acknowledgement to caller}
  * That they have been told of having a heart condition
  * Interest in hearing more and possibly participating in the study

Exclusion Criteria:

* Member had case management and this was closed within the 30 days prior to identification for the study
* End-of life, terminal cancer, end stage renal disease, hospice, late stage Alzheimer's disease, dementia, ventricular assist device, heart transplant or active in heart transplant program. Excluded diagnoses or conditions will be identified where it is evident through Aetna's Health Profile Data diagnoses in claims, or upon case management assessment.
* Chronic or ongoing intravenous heart failure medication
* Any response to Interactive Voice Response outreach call other than "Yes, I am interested"

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time to acute hospital admission | 6 months
  During the 6 month intervention period, it is expected that the time from entering the study until the first primary event (acute hospital admission, emergency room visit or death) will be, on average, longer for those using the Intel® Health Guide with case management (HG-CM) than for those in the routine case management (Case Management-Only Group). The primary measure to be compared across the study groups will be the unadjusted hazard ratio.
Acute Hospital Admission, Emergency Room Visit or Death | 6 months
  It is expected that the proportion of members with an inpatient acute admission, emergency room visit, or death in the intervention period and follow-up periods will be lower in the HG-CM Group than the Case Management-Only Group.

SECONDARY OUTCOMES:
Decrease the number of acute hospital admissions and emergency room visits | 6 months
  Number of acute hospital admissions and emergency room visits will decrease during the 6 month intervention period and the number during the 3 months after the intervention period
Number of Inpatient Hospital Days associated with Acute Admissions | 6 months
  Medicare members using the Intel® Health Guide are expected to have fewer Inpatient Acute Days in the intervention 6 months and during the 3 month follow-up period than do those in the Case Management-Only Group.
Cardiovascular Admissions Decreased | 6 months
  Number of members with a hospital admission or emergency room visit for a cardiovascular DRG diagnosis in the intervention 6 months or during the 3 months' follow-up period will decrease

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Wade, MD, Principal Investigator — Aetna, Inc.
Locations (1):
- Aetna, Princeton, New Jersey, United States